CLINICAL TRIAL: NCT01185041
Title: Effects of Oral L-citrulline/L-arginine in Watermelon on Central Blood Pressure and Arterial Stiffness in Individuals With Obesity-related High Blood Pressure
Brief Title: Watermelon Supplementation and Arterial Stiffness
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Associate Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RF02032
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Hypertension
Keywords: Arterial Stiffness; Wave Reflection; Watermelon Supplementation; Aortic Blood Pressure; Obesity
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maltodextrin (Placebo Comparator): 6g/day of placebo (maltodextrin)
  Interventions: Dietary Supplement: Watermelon Extract
- Watermelon (Experimental): (6g per day)containing L-citrulline/L-arginine (4/2 g)
  Interventions: Dietary Supplement: Watermelon Extract

INTERVENTIONS:
Dietary Supplement: Watermelon Extract — 6 weeks of watermelon extract taken in two doses of 3g each per day (6g per day)containing L-citrulline/L-arginine (4/2 g)
  Other Names: Watermelon extract from Milne fruit Products Inc

SUMMARY:
Increased abdominal obesity (waist circumference) and systolic blood pressure (BP) are main risk factors for the metabolic syndrome. Approximately 60% of adults in the United States are prehypertensive or hypertensive. Hypertension has been associated with abnormal endothelial and autonomic function, the two main mechanisms of BP regulation. Endothelial dysfunction, as a result of reduced NO (a vasodilator), and increased sympathetic nervous system activity contribute to arterial stiffness by enhancing the vasomotor tone. Because BP variations are sensed by baroreceptors in the wall of large arteries, increased stiffness of arteries may attenuate the control of BP by the autonomic nervous system leading to hypertension. High production of proinflammatory cytokines and low adiponectin (vascular protective molecule), are considered the underlying mechanisms leading to endothelial dysfunction and arterial stiffness. The recommended intervention for controlling BP in overweight/obese individuals with pre- and stage 1- hypertension is lifestyle modifications and not drug therapy. Among the dietary regimens that are reported to reduce BP is L-arginine, the substrate for endothelial NO production. Recently, oral L-citrulline has been shown to be more effective than L-arginine in improving circulating NO levels because is not affected by enzymatic degradation. Watermelon, the leading US melon crop, is one of the few natural foods rich in L-citrulline which is efficiently transformed to arginine in humans. The investigators long-term goal is to provide feasible and effective dietary ways to reduce cardiovascular risk factors in individuals with high abdominal fat and BP. The overall objective of this study is to bring forth evidence that watermelon supplementation will reduce BP and cardiovascular risk factors such as arterial stiffness, autonomic dysfunction and endothelial dysfunction. The investigators postulate that watermelon supplementation will reduce BP and arterial stiffness by enhancing endothelial function and reducing vascular inflammation. The findings of this study will provide a foundation for disseminating feasible, safe approaches for preventing and combating obesity-related hypertension at its early stage which does not require drug therapy.

DETAILED DESCRIPTION:
The purpose of the study is to examine the effect of 12 weeks of L-citrulline/L-arginine in the form of watermelon supplementation on arterial function and autonomic neural control of the heart rate and blood pressure in older overweight/obese men and women with pre- and stage 1- hypertension. The specific aims of the study are:

1. To investigate the extent to which daily consumption of watermelon supplementation containing L-citrulline/L-arginine (4/2 g) will reduce BP and arterial stiffness. This aim will examine the working hypothesis that watermelon supplementation will reduce BP and improve arterial function. This aim will be tested by measuring brachial and central (aortic and carotid) BP at rest and during physiological stress (head-up tilt test and cold pressor test), and by evaluating arterial stiffness using pulse wave velocity of the aorta and legs as primary variables.
2. To determine the effect of watermelon supplementation on endothelial function. There is evidence that watermelon improves endothelial function in rats. Hence, we postulate that watermelon in part exerts its vascular protective effects by modulating indices of endothelial function. This aim will be tested by measuring flow-mediated dilation using vascular ultrasound and circulating levels of vasodilators, vasoconstrictors, and markers of vascular inflammation (adiponectin, leptin, endothelin-1, angiotensin II, prostaglandin F2α, sVCAM-1, sICAM-1, and 8-isoprostane).
3. To determine whether watermelon supplementation will improve the autonomic control of BP and heart rate in individuals with high abdominal obesity and BP. There is evidence that food high in L-arginine improves baroreflex sensitivity (BRS) in individuals with pre-hypertension. This aim will examine the working hypothesis that watermelon will improve cardiovascular autonomic control of BP by measuring heart rate variability, BP variability and BRS at rest and during physiological stress as secondary variables.

ELIGIBILITY:
Inclusion Criteria:

* Thirty men and women 45-70 years of age
* BP between 120-159/80-99 mmHg
* Waist circumference >102 cm in men and > 80 cm in women

Exclusion Criteria:

* BP >160/100 mmHg
* Asthma
* Glaucoma
* Herpes simplex
* Uncontrolled diabetes
* Neurological disease
* Cardiovascular disease
* Inflammatory disease
* Kidney disease
* Hormone replacement therapy (HRT)
* Amino acid/vitamin supplementation\
* Corticosteroids or non-steroidal anti-inflammatory drugs
* Any drug known to affect BP or heart rate
* Glycemic control drugs
* Lipids reducing drugs
* Participants should not consume > 12 alcoholic drink/week
* Smokers
* Regular Exercisers (= 1.5 hour/week).

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 12 weeks
  By measuring brachial and central (aortic and carotid) BP at rest and during physiological stress (head-up tilt test and cold pressor test)

SECONDARY OUTCOMES:
Arterial Stiffness | 12 weeks
  Using pulse wave velocity of the aorta and legs.
Endothelial function | 12 weeks
  By measuring flow-mediated dilation using vascular ultrasound and circulating levels of vasodilators, vasoconstrictors, and markers of vascular inflammation (adiponectin, leptin, endothelin-1, angiotensin II, prostaglandin F2α, sVCAM-1, sICAM-1, and 8-isoprostane).
Autonomic control of BP | 12 weeks
  By measuring BP variability and BRS at rest and during physiological stress
Autonomic control of heart rate | 12 weeks
  By measuring heart rate variability at rest and during physiological stress

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, MD, PhD, Principal Investigator — The Florida State University
Locations (1):
- Cardiovascular Physiology Laboratory, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Figueroa A, Wong A, Kalfon R. Effects of watermelon supplementation on aortic hemodynamic responses to the cold pressor test in obese hypertensive adults. Am J Hypertens. 2014 Jul;27(7):899-906. doi: 10.1093/ajh/hpt295. Epub 2014 Feb 26. PMID 24572702